CLINICAL TRIAL: NCT01702558
Title: Phase I Study of the Combination of Trastuzumab Emtansine (T-DM1) and Capecitabine in HER2-Positive Metastatic Breast Cancer and HER2-Positive Locally Advanced/Metastatic Gastric Cancer Patients, Followed by a Randomized, Open-Label Phase II Study of Trastuzumab Emtansine and Capecitabine Versus Trastuzumab Emtansine Alone in HER2-Positive Metastatic Breast Cancer
Brief Title: A Combination Study of Kadcyla (Trastuzumab Emtansine) and Capecitabine in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Breast Cancer (mBC) or HER2-Positive Locally Advanced/Metastatic Gastric Cancer (LA/mGC)
Acronym: TRAXHER2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to terminate study after 70% of participants had experienced a progression-free survival event.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MO28230; 2012-001547-46 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — Capecitabine; Ado-Trastuzumab Emtansine

ARMS (4):
- Phase 1 (mBC) Cohort 1: T-DM1 + Capecitabine (Experimental): In Phase 1, Cohort 1 participants (with mBC) will receive trastuzumab emtansine (T-DM1) at a dose of 3.6 milligrams per kilogram (mg/kg) via intravenous (IV) infusion (on Day 1 [on Day 2 for Cycle 1] of each 21-day cycle) along with capecitabine at de-escalating dose levels (starting from 750 milligrams per meter squared [mg/m^2]) via tablet orally twice daily on Days 1-14 of each 21-day cycle until unacceptable toxicity, withdrawal of consent, disease progression (PD), death, or study end.
  Interventions: Drug: Capecitabine; Drug: Trastuzumab emtansine (T-DM1)
- Phase 1 (LA/mGC) Cohort 2: T-DM1 + Capecitabine (Experimental): In Phase 1, Cohort 2 participants (with LA/mGC) will receive trastuzumab emtansine at a dose of 2.4 mg/kg via IV infusion on Day 1 (on Day 2 of first week) of every week along with capecitabine at MTD (determined in Cohort 1) via tablet orally twice daily on Days 1-14 followed by a 7-day rest period, in each 21-day cycle until unacceptable toxicity, withdrawal of consent, PD, death, or study end.
  Interventions: Drug: Trastuzumab emtansine (T-DM1); Drug: Capecitabine
- Phase 2 (mBC): T-DM1 + Capecitabine (Active Comparator): In Phase 2, participants (with mBC) who will be randomized to this group, will receive trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion on Day 1 of each 21-day cycle along with capecitabine at MTD via tablet orally twice daily on Days 1-14 of each 21-day cycle until unacceptable toxicity, withdrawal of consent, PD, death, or study end.
  Interventions: Drug: Trastuzumab emtansine (T-DM1); Drug: Capecitabine
- Phase 2 (mBC): T-DM1 (Experimental): In Phase 2, participants (with mBC) who will be randomized to this group, will receive trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion on Day 1 of each 21-day cycle until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, or study end.
  Interventions: Drug: Trastuzumab emtansine (T-DM1)

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered at de-escalating doses (starting from 750 mg/m^2) to determine the MTD.
  Other Names: Xeloda
  Arms: Phase 1 (mBC) Cohort 1: T-DM1 + Capecitabine
Drug: Trastuzumab emtansine (T-DM1) — Trastuzumab emtansine will be administered at a dose of 3.6 mg/kg via IV infusion every 3 weeks.
  Other Names: Kadcyla,; RO5304020
  Arms: Phase 1 (mBC) Cohort 1: T-DM1 + Capecitabine; Phase 2 (mBC): T-DM1; Phase 2 (mBC): T-DM1 + Capecitabine
Drug: Trastuzumab emtansine (T-DM1) — Trastuzumab emtansine will be administered at a dose of 2.4 mg/kg via IV infusion every week.
  Other Names: Kadcyla,; RO5304020
  Arms: Phase 1 (LA/mGC) Cohort 2: T-DM1 + Capecitabine
Drug: Capecitabine — Capecitabine will be administered at the MTD determined in Cohort 1.
  Other Names: Xeloda
  Arms: Phase 1 (LA/mGC) Cohort 2: T-DM1 + Capecitabine; Phase 2 (mBC): T-DM1 + Capecitabine

SUMMARY:
This multicenter study will assess the maximum tolerated dose (MTD) of capecitabine in combination with Kadcyla (trastuzumab emtansine) in participants with HER2-positive mBC or HER2-positive LA/mGC using a Phase 1 design, followed by a randomized, open-label Phase 2 part to explore the efficacy and safety of the combination of Kadcyla and capecitabine compared with Kadcyla alone in participants with mBC. The anticipated time on study treatment is until disease progression, intolerable toxicity, withdrawal of consent, or study end.

ELIGIBILITY:
Inclusion Criteria:

Metastatic Breast Cancer

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate blood cell count
* Adequate liver, renal, and cardiac function
* Life expectancy greater than or equal to (>/=) 12 weeks
* Histologically or cytologically confirmed breast cancer
* Confirmed HER2-positive disease, defined as immunohistochemistry (IHC) 3+ or in situ hybridization (ISH)-positive
* mBC with at least one measurable lesion according to RECIST v1.1
* Disease progression on at least one prior regimen containing trastuzumab and chemotherapy either separately or in combination; participants may be eligible to receive study therapy in first-line setting if trastuzumab and chemotherapy were given in the neoadjuvant/adjuvant setting
* Participant must have recovered from previous treatments

Locally Advanced/Metastatic Gastric Cancer

* ECOG performance status of 0, 1, or 2
* Adequate blood cell count
* Adequate liver, renal, and cardiac function
* Life expectancy >/= 12 weeks
* Histologically or cytologically confirmed LA/mGC
* HER2-positive tumor (primary tumor or metastatic lesion), defined as either IHC 3+ or IHC 2+ and ISH-positive
* Inoperable LA/mGC

Exclusion Criteria:

Metastatic Breast Cancer

* Prior treatments before first study treatment:

  1. Investigational therapy within 28 days or 5 half-lives, whichever is longer
  2. Hormonal therapy within 14 days
  3. Trastuzumab within 21 days
* Prior treatment with trastuzumab emtansine or prior enrollment in a trastuzumab emtansine-containing study, regardless of whether the patient received trastuzumab emtansine
* Prior treatment with capecitabine
* History of severe or unexpected reactions to fluoropyrimidine or known hypersensitivity to fluorouracil
* Related capecitabine contraindications

  1. Treatment with sorivudine or chemically-related analogues
  2. Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
  3. Complete absence of dihydropyrimidine dehydrogenase (DPD) activity
* History of intolerance or hypersensitivity to trastuzumab or murine proteins or any product component
* History of exposure to high cumulative doses of anthracyclines
* Brain metastases that are symptomatic or require radiation, surgery, or steroid therapy to control symptoms within 28 days before study drug
* Current peripheral neuropathy of Grade >/=3
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome
* Current unstable ventricular arrhythmia requiring treatment
* History of symptomatic congestive heart failure (CHF)
* History of myocardial infarction or unstable angina within 6 months prior to study drug
* History of left ventricular ejection fraction (LVEF) less than (<) 40% or symptomatic CHF with previous trastuzumab treatment
* Severe dyspnea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy
* Clinically significant malabsorption syndrome or inability to take oral medication
* Current severe, uncontrolled systemic disease (such as clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during study treatment
* Current known active infection with human immunodeficiency virus (HIV) or hepatitis B or C
* Lapatinib within 14 days before study drug

Locally Advanced/Metastatic Gastric Cancer

* Same as above, with addition of previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- Argentina (2):
  - Fundacion Investigar, CABA
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Brazil (4):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Instituto Oncologico de Ribeirao Preto - INORP, Ribeirão Preto, São Paulo
  - Faculdade de Medicina de Sao Jose do Rio Preto - FAMERP*X*, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia, Canada
- France (5):
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Paoli Calmettes; Oncologie Medicale, Marseille
  - Institut Curie; Oncologie Medicale, Paris
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
- Germany (7):
  - Charité-Universitätsm. Berlin; Med. Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunolo., Berlin
  - Onkologische Schwerpunktpraxis Bielefeld; Haemotologie & Internistische onkologie, Bielefeld
  - Heinrich-Heine Universitätsklinik Düsseldorf, Düsseldorf
  - Klinik Fulda, Medizinisches Versorgungszentrum Osthessen GmbH, Fulda
  - Philipps-Universität Marburg; Klinik für Innere Med.; Schwerpunkt Hämatologie/Onkologie/Immunologie, Marburg
  - Klinikum rechts der Isar der TU München; III. Medizinischen Klinik (Hämatologie/Onkologie), München
  - Klinikum rechts der Isar der TU München; Klinik und Poliklinik für Frauenheilkunde, München
- Greece (3):
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Patras Medical Oncology, Pátrai
- Italy (4):
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE;U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Azienda usl 5 Di Pisa-Ospedale Di Pontedera;U.O. Oncologia, Pontedera, Tuscany
- Portugal (3):
  - Hospital da Luz; Departamento de Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Russia (6):
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Blokhin Cancer Research Center; Combined Treatment, Moscow
  - City Clinical Oncology Hospital, Moscow
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg
  - City Oncology Dispensary, Saint Petersburg
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia; Medical Oncology, Belgrade
  - Clinical Centre Nis, Clinic for Oncology, Niš
- Slovakia (2):
  - Narodny Onkologicky Ustav; Oddelenie klinickej onkologie A, Bratislava
  - Fakultna nemocnica Trencín; Onkologicke odd., Trenčín
- Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona, Spain

REFERENCES:
- [Derived] Cortes J, Dieras V, Lorenzen S, Montemurro F, Riera-Knorrenschild J, Thuss-Patience P, Allegrini G, De Laurentiis M, Lohrisch C, Oravcova E, Perez-Garcia JM, Ricci F, Sakaeva D, Serpanchy R, Sufliarsky J, Vidal M, Irahara N, Wohlfarth C, Aout M, Gelmon K. Efficacy and Safety of Trastuzumab Emtansine Plus Capecitabine vs Trastuzumab Emtansine Alone in Patients With Previously Treated ERBB2 (HER2)-Positive Metastatic Breast Cancer: A Phase 1 and Randomized Phase 2 Trial. JAMA Oncol. 2020 Aug 1;6(8):1203-1209. doi: 10.1001/jamaoncol.2020.1796. PMID 32584367

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 234 participants were screened, out of which, 182 participants were enrolled into the study. Out of the 182 enrolled participants, 3 participants were excluded from all safety and efficacy analyses because they did not sign correct Informed Consent Form (ICF).
Groups:
- Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape: In Phase 1, Cohort 1 participants (with mBC) received trastuzumab emtansine (T-DM1) at a dose of 3.6 milligrams per kilogram (mg/kg) via intravenous (IV) infusion (on Day 1 [on Day 2 for Cycle 1] of each 21-day cycle) along with capecitabine (Cape) at a dose level (DL) of 750 milligrams per meter squared (mg/m^2) via tablet orally twice daily on Days 1-14 of each 21-day cycle until unacceptable toxicity, withdrawal of consent, disease progression (PD), death, reasons deemed by the treating physician, or study termination by the sponsor.
- Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape: In Phase 1, Cohort 1 participants (with mBC) received trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion (on Day 1 [on Day 2 for Cycle 1] of each 21-day cycle) along with capecitabine at a dose level of 700 mg/m^2 via tablet orally twice daily on Days 1-14 of each 21-day cycle until unacceptable toxicity, withdrawal of consent, PD, death, reasons deemed by the treating physician, or study termination by the sponsor.
- Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape: In Phase 1, Cohort 2 participants (with LA/mGC) received trastuzumab emtansine at a dose of 2.4 mg/kg via IV infusion on Day 1 (Day 2 of first week) of every week along with capecitabine at a dose level of 700 mg/m^2 via tablet orally twice daily on Days 1-14 followed by a 7-day rest period, in each 21-day cycle until unacceptable toxicity, withdrawal of consent, PD, death, reasons deemed by the treating physician, or study termination by the sponsor.
- Phase 2 (mBC): T-DM1 + Cape: In Phase 2, participants (with mBC) who were randomized to this group received trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion on Day 1 of each 21-day cycle along with capecitabine at a dose level of 700 mg/m^2 via tablet orally twice daily on Days 1-14 of each 21-day cycle until unacceptable toxicity, withdrawal of consent, PD, death, reasons deemed by the treating physician, or study termination by the sponsor.
- Phase 2 (mBC): T-DM1: In Phase 2, participants (with mBC) who were randomized in this group received trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion on Day 1 of each 21-day cycle until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.
Period: Overall Study
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Started | 7 | 5 | 6 | 81 | 80
Completed | 3 | 1 | 1 | 34 | 38
Not Completed | 4 | 4 | 5 | 47 | 42
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 12 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 0
Not completed — Death | 4 | 3 | 3 | 16 | 20
Not completed — Safety Follow-Up less than 3 Months | 0 | 0 | 2 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 16 | 17

BASELINE CHARACTERISTICS:
Population: Safety population: Participants who received >/=1 dose of study drug, analyzed as per actual treatment received. In Phase 2, of 161 participants, 1 was randomized in error(received no treatment) and was excluded from safety analysis and 1 who was randomized to T-DM1 alone Arm received Capecitabine throughout study and was counted in T-DM1+Cape Arm.
Groups:
- Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape: In Phase 1, Cohort 1 participants (with mBC) received trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion (on Day 1 [on Day 2 for Cycle 1] of each 21-day cycle) along with capecitabine at a dose level of 750 mg/m^2 via tablet orally twice daily on Days 1-14 of each 21-day cycle until unacceptable toxicity, withdrawal of consent, PD, death, reasons deemed by the treating physician, or study termination by the sponsor.
- Phase 2 (mBC): T-DM1: In Phase 2, participants (with mBC) who were randomized to this group received trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion on Day 1 of each 21-day cycle until investigator-assessed PD, unacceptable toxicity, withdrawal of consent, death, reasons deemed by the treating physician, or study termination by the Sponsor.
- Total: Total of all reporting groups
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1 | Total
Number analyzed (Participants) | 7 | 5 | 6 | 82 | 78 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.75) | 50.8 (7.76) | 60.0 (7.40) | 53.3 (11.69) | 52.6 (11.19) | 53.2 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 0 | 81 | 78 | 170
  Male | 1 | 0 | 6 | 1 | 0 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian | 6 | 4 | 6 | 71 | 65 | 152
  Race: N/A (as per local regulation) | 1 | 1 | 0 | 10 | 7 | 19
  Race: Black | 0 | 0 | 0 | 0 | 2 | 2
  Race: Asian | 0 | 0 | 0 | 1 | 1 | 2
  Race: Mixed | 0 | 0 | 0 | 0 | 3 | 3
  Ethnicity: Hispanic/Latino | 0 | 1 | 0 | 5 | 10 | 16
  Ethnicity: Chinese | 0 | 0 | 0 | 1 | 0 | 1
  Ethnicity: Other | 6 | 0 | 0 | 39 | 35 | 80
  Ethnicity: N/A (as per local regulation) | 1 | 1 | 6 | 32 | 29 | 69
  Ethnicity: Unknown | 0 | 2 | 0 | 5 | 4 | 11
  Ethnicity: Mixed | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 (mBC): Percentage of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any one of the following study treatment related toxicities: Uncomplicated Grade 4 thrombocytopenia that does not recover before Day 21; thrombocytopenia complicated with clinically significant bleeding requiring medical intervention; Grade 4 neutropenia lasting more than (>) 7 consecutive days; febrile neutropenia with absolute neutrophil count (ANC) less than (<) 1000 cells/millimeter cube (mm^3); Grade greater than or equal to (>/=) 3 diarrhea or Grade 3 hand-foot syndrome (in absence of dihydropyrimidine dehydrogenase [DPD] deficiency only for DL 1); any other Grade >/=3 toxicity prohibiting start of Cycle 2; Grade 2 toxicity requiring treatment interruption for >14 days (>7 days for DL 1); for DL -1 only: <14 full doses of capecitabine; Cycle 2 dose level <100 percent (%).
Time Frame: Continuously during Cycle 1 (up to 3 weeks)
Population: Analysis was performed on Phase 1 DLT-evaluable population for mBC cohort, which included all enrolled and treated mBC participants who did not experience any major protocol deviation and completed Cycle 1.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6 | 5
percentage of participants | 33.3 | 0.0

2. Primary Outcome: Phase 1 (mBC): Maximum Tolerated Dose (MTD) of Capecitabine When Combined With Trastuzumab Emtansine (3.6 mg/kg Every 3 Weeks)
Description: MTD was defined as the dose level for which the probability of DLT is equal to a protocol-specified target probability. A DLT was defined as any one of the following study treatment related toxicities: Uncomplicated Grade 4 thrombocytopenia that does not recover before Day 21; thrombocytopenia complicated with clinically significant bleeding requiring medical intervention; Grade 4 neutropenia lasting >7 consecutive days; febrile neutropenia with ANC <1000 cells/mm^3; Grade >/=3 diarrhea or Grade 3 hand-foot syndrome (in absence of DPD deficiency only for DL 1); any other Grade >/=3 toxicity prohibiting start of Cycle 2; Grade 2 toxicity requiring treatment interruption for >14 days (>7 days for DL 1); for DL -1 only: <14 full doses of capecitabine; Cycle 2 dose level <100%.
Time Frame: Continuously during Cycle 1 (up to 3 weeks)
Population: Analysis was performed on Phase 1 DLT-evaluable population for mBC cohort.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1 (mBC) Cohort 1: T-DM1 + Cape: In Phase 1, Cohort 1 participants (with mBC) received trastuzumab emtansine at a dose of 3.6 mg/kg via IV infusion (on Day 1 [on Day 2 for Cycle 1] of each 21-day cycle) along with capecitabine at a dose level of 700 or 750 mg/m^2 via tablet orally twice daily on Days 1-14 of each 21-day cycle until unacceptable toxicity, withdrawal of consent, PD, death, reasons deemed by the treating physician, or study termination by the sponsor.
Arm/Group | Phase 1 (mBC) Cohort 1: T-DM1 + Cape
Number analyzed (Participants) | 11
mg/m^2 | 700

3. Primary Outcome: Phase 2 (mBC): Percentage of Participants With Best Overall Response (BOR) as Assessed by the Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Tumor response was assessed by the investigator according to RECIST v1.1. BOR was defined as percentage of participants with a complete response (CR) or partial response (PR) that was confirmed by repeat assessments >/=4 weeks after initial documentation. CR was defined as the disappearance of all target lesions (TLs) and non-TLs; short axis (SA) reduction to <10 millimeters (mm) for nodal TLs/non-TLs; and no new lesions. PR was defined as >/=30% decrease in sum of diameters (SoD) of TLs, taking as reference the baseline SoD; no progression in non-TLs; and no new lesions. The 90% confidence Interval (CI) was computed using Clopper-Pearson approach.
Time Frame: Baseline until CR/PR, consent withdrawal, or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on Intent-to-Treat (ITT) Population, which included all participants in the randomized Phase 2 part of the study. Participants were analyzed as per the initial randomization. Participants without tumor assessment after start of study treatment were considered as non-responders.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
percentage of participants | 44.4 [35.0 to 54.2] | 36.3 [27.3 to 46.0]
Statistical Analysis 1: Comparison: Phase 2 (mBC): T-DM1 + Cape vs Phase 2 (mBC): T-DM1; Test type: Superiority; p = 0.336, Fisher Exact; Difference in Response Rates = 8.2, 90% CI 2-sided [-4.5 to 20.9] — 90% CI was estimated using Hauck-Anderson approach

4. Primary Outcome: Phase 1 (LA/mGC): Percentage of Participants With DLTs
Description: A DLT was defined as any one of the following study treatment related toxicities: Uncomplicated Grade 4 thrombocytopenia that does not recover before Day 21; thrombocytopenia complicated with clinically significant bleeding requiring medical intervention; Grade 4 neutropenia lasting >7 consecutive days; febrile neutropenia with ANC <1000 cells/mm^3; Grade >/=3 diarrhea or Grade 3 hand-foot syndrome; any other Grade >/=3 toxicity prohibiting start of Cycle 2; Grade 2 toxicity requiring treatment interruption for >14 days; <14 full doses of capecitabine; Cycle 2 dose level <100%.
Time Frame: Continuously during 3 weeks
Population: Analysis was performed on Phase 1 DLT-evaluable population for LA/mGC cohort, which included all enrolled and treated LA/mGC participants who did not experience any major protocol deviation and completed Cycle 1.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
percentage of participants | 0.0

5. Primary Outcome: Phase 1 (LA/mGC): MTD of Capecitabine When Combined With Trastuzumab Emtansine (2.4 mg/kg QW)
Description: MTD was defined as the dose level for which the probability of DLT is equal to a protocol-specified target probability. A DLT was defined as any one of the following study treatment related toxicities: Uncomplicated Grade 4 thrombocytopenia that does not recover before Day 21; thrombocytopenia complicated with clinically significant bleeding requiring medical intervention; Grade 4 neutropenia lasting >7 consecutive days; febrile neutropenia with ANC <1000 cells/mm^3; Grade >/=3 diarrhea or Grade 3 hand-foot syndrome; any other Grade >/=3 toxicity prohibiting start of Cycle 2; Grade 2 toxicity requiring treatment interruption for >14 days; <14 full doses of capecitabine; Cycle 2 dose level <100%.
Time Frame: Continuously during 3 weeks
Population: Analysis was performed on Phase 1 DLT-evaluable population for LA/mGC cohort.
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
mg/m^2 | 700

6. Secondary Outcome: Phase 1 (mBC): Percentage of Participants With BOR as Assessed by the Investigator According to RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. BOR in Phase 1 was defined as percentage of participants with a CR or PR. CR was defined as the disappearance of all TLs and non-TLs; SA reduction to <10 mm for nodal TLs/non-TLs; and no new lesions. PR was defined as >/=30% decrease in SoD of TLs, taking as reference the baseline SoD; no progression in non-TLs; and no new lesions.
Time Frame: Baseline until CR/PR, consent withdrawal, or study end whichever occurred first (up to approximately 3.5 years overall)
Population: Analysis was performed on Phase 1 DLT-evaluable population for mBC cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6 | 5
percentage of participants | 83.3 | 100.0

7. Secondary Outcome: Phase 1 (mBC): Serum Concentration of Trastuzumab Emtansine
Time Frame: Pre-trastuzumab emtansine dose (0 hour [h]) on Day 1 Cycle 2; 15-30 minutes (min) after end of trastuzumab emtansine infusion (maximum infusion duration = 90 min) on Day 2 Cycle 1 and Day 1 Cycle 2 (cycle length=21 days)
Population: Phase 1 pharmacokinetic (PK) analysis population for mBC cohort; included all mBC participants receiving at least one dose of study medication during Phase 1 and had at least one reported serum/plasma result for PK. The PK analysis in mBC cohort included 1 patient who was excluded from the main safety and efficacy analyses due to ICF issues.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
micrograms per milliliter (mcg/mL)
  Cycle 1, Post-dose | 81.3 (13.3) | 78.6 (14.6)
  Cycle 2, Pre-dose | 1.17 (1.25) | 2.1 (1.49)
  Cycle 2, Post-dose | 70.5 (13.3) | 78.5 (14.9)

8. Secondary Outcome: Phase 1 (mBC): Serum Concentration of Trastuzumab
Description: Trastuzumab was derived from trastuzumab emtansine.
Time Frame: Pre-trastuzumab emtansine dose (0 h) on Day 1 Cycle 2; 15-30 min after end of trastuzumab emtansine infusion (maximum infusion duration = 90 min) on Day 2 Cycle 1 and Day 1 Cycle 2 (cycle length=21 days)
Population: Analysis was performed on Phase 1 PK analysis population for mBC cohort. The PK analysis in the mBC cohort included 1 patient who was excluded from the main safety and efficacy analyses due to ICF issues.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
mcg/mL
  Cycle 1, Post-dose | 89.1 (24.37) | 92.9 (22.13)
  Cycle 2, Pre-dose | 11.8 (13.28) | 14.0 (12.53)
  Cycle 2, Post-dose | 74.8 (18.89) | 94.7 (24.60)

9. Secondary Outcome: Phase 1 (mBC): Maximum Observed Plasma Concentration (Cmax) of Capecitabine
Description: Cmax for Capecitabine was estimated from plasma concentration versus time data using non-compartmental methods of analysis. Reported dispersion values are for percent coefficient of variation (CV%) and not for standard deviation.
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
nanograms per milliliter (ng/mL) | 2990 (38.4) | 5652 (91.1)

10. Secondary Outcome: Phase 1 (mBC): Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC[0-inf]) of Capecitabine
Description: AUC(0-inf) is the measure of total drug exposure and is dependent on the total amount of drug absorbed. AUC(0-inf) for capecitabine was estimated from plasma concentration versus time data using non-compartmental methods of analysis. Reported dispersion values are for CV% and not for standard deviation.
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
hours*nanograms per milliliter (h*ng/mL) | 3973 (38.0) | 5440 (57.7)

11. Secondary Outcome: Phase 1 (mBC): Plasma Terminal Half-Life (t1/2) of Capecitabine
Description: Plasma terminal half-life is the time measured for the plasma drug concentration to decrease by one half during the elimination phase of the drug. t1/2 for capecitabine was estimated from plasma concentration versus time data using non-compartmental methods of analysis. Reported dispersion values are for CV% and not for standard deviation.
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
hours | 0.70 (131.9) | 0.39 (38.8)

12. Secondary Outcome: Phase 1 (mBC): Cmax of 5-Fluorouracil (Metabolite of Capecitabine)
Description: 5-fluorouracil is a metabolite of capecitabine. Cmax for 5-fluorouracil was estimated from plasma concentration versus time data using non-compartmental methods of analysis. Reported dispersion values are for CV% and not for standard deviation.
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
ng/mL | 148 (49.9) | 143 (45.6)

13. Secondary Outcome: Phase 1 (mBC): AUC(0-inf) of 5-Fluorouracil (Metabolite of Capecitabine)
Description: 5-fluorouracil is a metabolite of capecitabine. AUC(0-inf) is the measure of total drug exposure and is dependent on the total amount of drug absorbed. AUC(0-inf) for 5-fluorouracil was estimated from plasma concentration versus time data using non-compartmental methods of analysis. Reported dispersion values are for CV% and not for standard deviation.
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
h*ng/mL | 257 (49.9) | 244 (38.2)

14. Secondary Outcome: Phase 1 (mBC): t1/2 of 5-Fluorouracil (Metabolite of Capecitabine)
Description: 5-fluorouracil is a metabolite of capecitabine. Plasma terminal half-life is the time measured for the plasma drug concentration to decrease by one half during the elimination phase of the drug. t1/2 for 5-fluorouracil was estimated from plasma concentration versus time data using non-compartmental methods of analysis. Reported dispersion values are for CV% and not for standard deviation.
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 7 | 6
hours | 0.63 (39.5) | 0.64 (18.3)

15. Secondary Outcome: Phase 2 (mBC): Time to Response (TTR) as Assessed by the Investigator According to RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. TTR was defined as the time (in months) from randomization to first documentation of confirmed PR or CR (whichever occurred first). CR was defined as the disappearance of all TLs and non-TLs; SA reduction to <10 mm for nodal TLs/non-TLs; and no new lesions. PR was defined as >/=30% decrease in SoD of TLs, taking as reference the baseline SoD; no progression in non-TLs; and no new lesions.
Time Frame: Baseline until first documentation of confirmed PR or CR, whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population. Only participants with a BOR of CR or PR were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 36 | 29
months | 2.10 [1.2 to 10.8] | 2.10 [1.9 to 8.0]

16. Secondary Outcome: Phase 2 (mBC): Duration of Response (DoR) as Assessed by the Investigator According to RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. DoR was defined as the time (in months) from the date of first recorded PR/CR until the date of PD or death from any cause. CR: the disappearance of all TLs and non-TLs; SA reduction to <10 mm for nodal TLs/non-TLs; and no new lesions. PR: >/=30% decrease in SoD of TLs, taking as reference the baseline SoD; no progression in non-TLs; and no new lesions. PD: >/=20% relative increase with >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-TLs. Participants with no documented PD after CR/PR were censored at the time of last tumor assessment. Participants without post-baseline tumor assessment were censored at randomization plus 1 day. The median DOR and 90% CI were estimated using Kaplan-Meier method.
Time Frame: From the documentation of response until PD, death, consent withdrawal, or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population. Only participants with a BOR of CR or PR were included in the analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 36 | 29
months | 11.30 [8.61 to NA] — Upper limit of 90% CI could not be calculated due to insufficient number of participants who had an event. | 12.22 [8.84 to 15.97]

17. Secondary Outcome: Phase 2 (mBC): Percentage of Participants With PD as Assessed by the Investigator According to RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. PD was defined as >/=20% relative increase with >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-TLs.
Time Frame: Baseline until PD, consent withdrawal, or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
percentage of participants | 64.2 | 70.0

18. Secondary Outcome: Phase 2 (mBC): Time to Progression (TTP) as Assessed by the Investigator According to RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. TTP was defined as the time (in months) from randomization to the first occurrence of PD. PD was defined as >/=20% relative increase with >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-TLs. Participants with no documented PD at the time of study end (including participants who died before PD) or who were lost to follow-up were censored on the date of the last tumor assessment. The median TTP and 90% CI was estimated using Kaplan-Meier method.
Time Frame: Baseline until PD, consent withdrawal, or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
months | 10.38 [7.85 to 12.91] | 10.32 [7.56 to 13.27]

19. Secondary Outcome: Phase 2 (mBC): Percentage of Participants With Treatment Failure as Assessed by the Investigator According to RECIST v1.1
Description: Treatment failure was defined as occurrence of any of the following event while on treatment: PD, death, withdrawal due to adverse event (AE) or laboratory abnormality, or refusal of treatment. PD as assessed by the investigator according to RECIST v1.1 was defined as >/=20% relative increase with >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-TLs.
Time Frame: Baseline until treatment failure, consent withdrawal, or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
percentage of participants | 77.8 | 83.8

20. Secondary Outcome: Phase 2 (mBC): Time to Treatment Failure (TTF) as Assessed by the Investigator According to RECIST v1.1
Description: TTF was defined as the time (in months) from randomization until treatment failure (PD, death, withdrawal due to AE or laboratory abnormality, or refusal of treatment). PD as assessed by the investigator according to RECIST v1.1 was defined as >/=20% relative increase with >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-TLs. Participants who did not experience any of the above events while on study were censored on the date of their last tumor assessment. The median TTF and 90% CI was estimated using Kaplan-Meier method.
Time Frame: as for outcome 19
Population: Analysis was performed on ITT Population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
months | 9.86 [7.62 to 10.68] | 7.66 [6.54 to 10.68]

21. Secondary Outcome: Phase 2 (mBC): Percentage of Participants With PD as Assessed by the Investigator According to RECIST v1.1 or Death From Any Cause
Description: as for outcome 17
Time Frame: Baseline until PD, death from any cause, consent withdrawal, or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
percentage of participants | 67.9 | 73.8

22. Secondary Outcome: Phase 2 (mBC): Progression-Free Survival (PFS) as Assessed by the Investigator According to RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. PFS was defined as the time (in months) from randomization until the first documented PD or death from any cause, whichever occurred first. PD was defined as >/=20% relative increase with >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-TLs. Participants with no PFS events were censored on the date of the last tumor assessment. Participants without post-baseline tumor assessment were censored at randomization plus 1 day. The median PFS and 90% CI was estimated using Kaplan-Meier method.
Time Frame: as for outcome 21
Population: Analysis was performed on ITT Population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
months | 10.15 [7.85 to 12.55] | 9.82 [7.46 to 13.08]

23. Secondary Outcome: Phase 2 (mBC): Percentage of Participants With Clinical Benefit as Assessed by the Investigator According to RECIST v1.1
Description: The clinical benefit was defined as a confirmed response of CR, PR, or stable disease (SD) that lasted for at least 6 months. Tumor response was assessed by the investigator according to RECIST v1.1. CR: the disappearance of all TLs and non-TLs; SA reduction to <10 mm for nodal TLs/non-TLs; and no new lesions. PR: >/=30% decrease in SoD of TLs, taking as reference the baseline SoD; no progression in non-TLs; and no new lesions. PD: >/=20% relative increase with >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-TLs. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SoD on study. The 90% CI was computed using Clopper-Pearson approach.
Time Frame: Baseline until clinical benefit response, consent withdrawal, or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
percentage of participants | 66.7 [57.1 to 75.3] | 62.5 [52.7 to 71.6]

24. Secondary Outcome: Phase 2 (mBC): Percentage of Participants Who Died of Any Cause
Time Frame: Baseline until death or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
percentage of participants | 22.2 | 26.3

25. Secondary Outcome: Phase 2 (mBC): Overall Survival (OS)
Description: OS was defined as the time (in months) from randomization until death from any cause. Participants who were alive at the time of data cut-off were censored on the date of the last follow-up assessment. Participants who were lost to follow-up were censored as having no event (alive) on the date of last contact. The median OS and 90% CI was estimated using Kaplan-Meier method, which use the patients at risk as denominator rather than the whole number of patients.
Time Frame: Baseline until death or study end whichever occurred first (up to approximately 2.5 years overall)
Population: Analysis was performed on ITT Population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
Number analyzed (Participants) | 81 | 80
months | NA [NA to NA] — Median and 90% CI could not be calculated due to insufficient number of participants who had an event. | 24.71 [24.28 to NA] — Upper limit of 90% CI could not be calculated due to insufficient number of participants who had an event.

26. Secondary Outcome: Phase 1 (LA/mGC): Percentage of Participants With BOR as Assessed by the Investigator According to RECIST v1.1
Description: as for outcome 6
Time Frame: Baseline until CR/PR, consent withdrawal, or study end whichever occurred first (up to approximately 1.5 years overall)
Population: Analysis was performed on Phase 1 DLT-evaluable population for LA/mGC cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
percentage of participants | 83.3

27. Secondary Outcome: Phase 1 (LA/mGC): Serum Concentration of Trastuzumab Emtansine
Time Frame: as for outcome 8
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
mcg/mL
  Cycle 1, Post-dose | 30.1 (14.5)
  Cycle 2, Pre-dose | 10.1 (5.85)
  Cycle 2, Post-dose | 46.4 (7.74)

28. Secondary Outcome: Phase 1 (LA/mGC): Serum Concentration of Trastuzumab
Description: Trastuzumab was derived from trastuzumab emtansine.
Time Frame: as for outcome 8
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
mcg/mL
  Cycle 1, Post-dose | 33.1 (15.98)
  Cycle 2, Pre-dose | 18.5 (7.57)
  Cycle 2, Post-dose | 57.6 (13.55)

29. Secondary Outcome: Phase 1 (LA/mGC): Cmax of Capecitabine
Description: Cmax for capecitabine was estimated from plasma concentration versus time data using non-compartmental methods of analysis. Reported dispersion values are for CV% and not for standard deviation.
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
ng/mL | 4925 (36.3)

30. Secondary Outcome: Phase 1 (LA/mGC): AUC(0-inf) of Capecitabine
Description: as for outcome 10
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
h*ng/mL | 5131 (24.6)

31. Secondary Outcome: Phase 1 (LA/mGC): t1/2 of Capecitabine
Description: as for outcome 11
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
hours | 0.65 (34.5)

32. Secondary Outcome: Phase 1 (LA/mGC): Cmax of 5-Fluorouracil (Metabolite of Capecitabine)
Description: as for outcome 12
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
ng/mL | 137 (24.3)

33. Secondary Outcome: Phase 1 (LA/mGC): AUC(0-inf) of 5-Fluorouracil (Metabolite of Capecitabine)
Description: as for outcome 13
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
h*ng/mL | 213 (16.2)

34. Secondary Outcome: Phase 1 (LA/mGC): t1/2 of 5-Fluorouracil (Metabolite of Capecitabine)
Description: as for outcome 14
Time Frame: Pre-capecitabine dose (0 h) and 0.5, 1, 1.5, 2, 2.5, 4, and 6 h post-capecitabine dose on Day 1 Cycle 1
Population: Analysis was performed on Phase 1 PK analysis population for LA/mGC cohort.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape
Number analyzed (Participants) | 6
hours | 0.83 (17.0)

ADVERSE EVENTS:
Time Frame: Phase 1: Baseline up to 42 days after last dose (up to approximately 1.5 years overall); Phase 2: Baseline up to 42 days after last dose (up to approximately 2.5 years overall)
Description: Safety population included all participants who received >/=1 dose of study drug. Participants were analyzed as per actual treatment received. In Phase 2, out of 161 participants, 1 participant was randomized in error (did not receive any treatment) and was excluded from safety analysis and 1 participant who was randomized to T-DM1 alone Arm received Capecitabine throughout study and was counted in T-DM1+Cape Arm.
Arm/Group | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape | Phase 2 (mBC): T-DM1 + Cape | Phase 2 (mBC): T-DM1
All-Cause Mortality (participants affected / at risk) | 4/7 | 3/5 | 3/6 | 18/82 | 21/78
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/5 | 4/6 | 11/82 | 10/78
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 6/6 | 75/82 | 64/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape (N=7) | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape (N=5) | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape (N=6) | Phase 2 (mBC): T-DM1 + Cape (N=82) | Phase 2 (mBC): T-DM1 (N=78)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Tumour excision (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (mBC) Cohort 1 (DL 1): T-DM1 + Cape (N=7) | Phase 1 (mBC) Cohort 1 (DL -1): T-DM1 + Cape (N=5) | Phase 1 (LA/mGC) Cohort 2 (DL -1): T-DM1 + Cape (N=6) | Phase 2 (mBC): T-DM1 + Cape (N=82) | Phase 2 (mBC): T-DM1 (N=78)
Nausea (Gastrointestinal disorders) | 3 | 4 | 3 | 27 | 18
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 7 | 7
Constipation (Gastrointestinal disorders) | 3 | 4 | 4 | 8 | 8
Gingival bleeding (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 16 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 1 | 6 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 6
Toothache (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 7 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 11 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 5 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 4 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 4 | 10 | 11
Asthenia (General disorders) | 3 | 1 | 0 | 17 | 15
Chills (General disorders) | 2 | 1 | 0 | 1 | 5
Gait disturbance (General disorders) | 1 | 2 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 13 | 15
Mucosal inflammation (General disorders) | 2 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 3 | 4
Influenza like illness (General disorders) | 0 | 1 | 2 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 1 | 0 | 0 | 0
Mucosal dryness (General disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 0 | 8 | 5
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 0 | 2 | 4
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 15 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 5 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 17 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 5
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 1 | 1 | 4
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1 | 27 | 31
Platelet count decreased (Investigations) | 4 | 0 | 0 | 12 | 13
Alanine aminotransferase increased (Investigations) | 4 | 0 | 1 | 20 | 24
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 6 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 2 | 9 | 10
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 8 | 16
Aspartate aminotransferase (Investigations) | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 10 | 11
Cell death (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 1 | 1 | 6 | 3
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0 | 0
Blindness (Eye disorders) | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Pterygium (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal ischaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 0 | 35 | 21
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 13 | 6
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 4 | 9 | 13
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Bloody discharge (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Skin lesion excision (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 5
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 5 | 15
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 4
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Spider naevus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Tumour excision (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 5 | 1
Liver palpable (Investigations) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 5

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate the study after 70% of participants had experienced a PFS event. Participants were allowed to continue treatment by enrolling into study NCT00781612 or by moving to commercial drug, depending on their country.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-03-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT01702558/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT01702558/SAP_001.pdf